CLINICAL TRIAL: NCT02798263
Title: Randomized Clinical Trials of Acupuncture Effectiveness in the Rehabilitation of Women Under the Physical and Functional Dysfunction to Surgical Treatment of Breast Cancer
Brief Title: Breast Cancer Rehabilitation With Acupuncture and Physical Therapy Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Gil Facina, Doctor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUSaoPaulo PT 4
Record Dates: First submitted 2016-05-16; First posted 2016-06-14 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I kinesiotherapy (Experimental): Treated with standard therapeutic exercise, pre-defined, based on stretching the neck muscles, shoulder girdle and upper limb exercises for ADM lasting 30 minutes
  Interventions: Other: Kinesiotherapy
- : Group II Acupuncture (Experimental): Treated with 30 minutes of classical acupuncture using predefined points
  Interventions: Other: Acupuncture
- Group III Stiper (Experimental): They will be used the same acupuncture points of the group II, but using the needles in place Stiper®
  Interventions: Other: Stiper

INTERVENTIONS:
Other: Kinesiotherapy — Compare the standard treatment of pain, by kinesiotherapy versus acupuncture and Stiper.Standard therapeutic exercise, pre-defined, based on stretching the neck muscles, shoulder girdle and upper limb exercises for ADM lasting 30 minutes.
  Arms: Group I kinesiotherapy
Other: Acupuncture — 30 minutes of classical acupuncture using predefined points.
  Arms: : Group II Acupuncture
Other: Stiper — They will be used the same acupuncture points of the group II, but using the needles in place Stiper.
  Arms: Group III Stiper

SUMMARY:
The pain is very common complaint, and the neck is one of the most affected spots, mainly due to muscle contracture of the cervical and scapular region, triggered by emotional stress associated with muscle retraction involved resulting from postoperative scarring or post-radiotherapy.O fear fibrosis move the limb and inactivity postoperative lead to gradual impairment of muscle strength and flexibility, and loss of ADM, which also predisposes to the appearance of pain.

Goals Study the effectiveness of acupuncture in rehabilitation of physical and functional disorders of women undergoing surgery for breast cancer.

1. Presence of pain by Visual Analog Scale of Pain (VAS).
2. Shoulder Range of Motion (ROM) by active goniometry of flexion movements, extension, adduction, abduction, internal rotation and external rotation
3. lymphedema presence through top member perimetry.
4. upper limb function through the DASH questionnaire.
5. Depressive symptoms through BECK questionnaire.
6. Quality of life through the EORTC questionnaire.
7. Muscle strength of flexion, extension, adduction, abduction, internal rotation and shoulder external rotation with the Hand Held Dynamometer 01,163 model of Lafayette Instrument Company.

Patients will be divided into three randomized groups with 30 patients per group, who will receive weekly treatment for 10 weeks, and the group I treated with standard therapeutic exercise, pre-defined, based on stretching the neck muscles, shoulder girdle and exercises for ADM upper limb lasting 30 minutes; group II is treated com30 minutes classical acupuncture using pre-defined spots, and finally, grupoIII be used in the same acupuncture points of the group II, but using the Stiper® in place of the needles. If the patients in groups II and III still of pain at the end of 10 sessions will be treated complementarily with kinesiotherapy.

DETAILED DESCRIPTION:
Objectives General Study the effectiveness of acupuncture in rehabilitation of physical and functional disorders of women undergoing surgery for breast cancer.

Specific

To evaluate the (the):

1. Presence of pain by Visual Analog Scale of Pain (VAS).
2. Shoulder Range of Motion (ROM) by active goniometry of flexion movements, extension, adduction, abduction, internal rotation and external rotation
3. lymphedema presence through top member perimetry.
4. upper limb function through the DASH questionnaire.
5. Depressive symptoms through BECK questionnaire.
6. Quality of life through the EORTC questionnaire.
7. Muscle strength of flexion, extension, adduction, abduction, internal rotation and shoulder external rotation with the Hand Held Dynamometer 01,163 model of Lafayette Instrument Company.

rationale The increased incidence of breast cancer and successful treatment result in greater survival. These patients may have chronic condition of pain in the area of the shoulder girdle and upper limb, including the thoracic and cervical spine. Knowing that in our previous project in which the group treated only with kinesiotherapy showed good results and when joined acupuncture no superiority, the investigators created new research study in order to determine whether acupuncture and Stiper® in isolated groups, would present equivalence results when compared to kinesiotherapy.The investigators propose then treat with acupuncture and analyze the rehabilitation of these patients.

methodology This study will be performed at the Clinic of the Department of Mastology the Department of Gynecology, Federal University of São Paulo (UNIFESP) - Paulista School of Medicine (EPM). Patients will be recruited, selected and informed about the study objectives, relevance, activities to be developed and the possibility of improvement, as well as answer your questions and concerns about the disease. Later the patients who wish to participate in the study protocol will sign a consent form and specific savy for this project.

ELIGIBILITY:
Inclusion Criteria:

* Underwent surgical treatment of breast cancer, radical or conservative, and exhibiting pain in the region of the shoulder girdle and upper limb, including thoracic and cervical spine after three months of surgery
* Patients should be older than 18 years
* Level of pain ≥ 3 on the Visual Analogue Scale (VAS)

Exclusion Criteria:

* Bilateral breast surgery
* Metastatic disease
* Vascular disorders and tactile sensitivity, with diabetes mellitus type I and II and decompensated with lower education level than four years

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Presence of pain | four years
  Presence of pain by Visual Analog Scale of Pain (VAS).

SECONDARY OUTCOMES:
shoulder range of motion | four years
  Shoulder range of motion by active goniometry of flexion movements, extension, adduction, abduction, internal rotation and external rotation in degrees
lymphedema presence | four years
  lymphedema presence through top member perimetry(centimeters).
upper limb function | four years
  upper limb function through the DASH questionnaire.
depressive symptoms | four years
  Depressive symptoms through BECK questionnaire.
quality of life of patients after breast cancer surgery | four years
  Quality of life through the EORTC questionnaire.
muscle strength | four years
  Muscle strength of flexion, extension, adduction, abduction, internal rotation and shoulder external rotation with the Hand Held Dynamometer 01,163 model of Lafayette Instrument Company(Kg).

CONTACTS AND LOCATIONS:
Locations (1):
- University Federal of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No